CLINICAL TRIAL: NCT00381420
Title: A Canadian Multi-Center, Randomized, Double-Blind Study of the Sirolimus-Coated BX Velocity Balloon-Expandable Stent in the Treatment of Patients With de Novo Coronary Artery Lesions.
Brief Title: The Study of the BX Velocity Stent in the Treatment of De Novo Artery Lesions.
Acronym: C-SIRIUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01-6307
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sirolimus-coated Bx Velocity stent
  Interventions: Device: drug-eluting stent
- 2 (Active Comparator): uncoated Bx Velocity stent
  Interventions: Device: bare-metal stent

INTERVENTIONS:
Device: drug-eluting stent — sirolimus-coated Bx VELOCITY Balloon-Expandable Stent
  Arms: 1
Device: bare-metal stent — un-coated Bx VELOCITY Stent
  Arms: 2

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus-coated Bx VELOCITY™ stent in maintaining minimum lumen diameter in de novo native coronary artery lesions as compared to the uncoated Bx VELOCITY™ balloon-expandable stent. Both stents are mounted on the Raptor® Stent Delivery Systems.

The secondary objective is to assess cost-effectiveness expressed in incremental cost/life year gained or cost/quality adjusted life year gained at different time points (8 months, 1 year, 3 and 5 years).

DETAILED DESCRIPTION:
This is a multicenter ,prospective, randomized double blind study. This study has a 2-arm design assessing the safety and effectiveness of the sirolimus-coated Bx VELOCITY™ stent to the uncoated Bx VELOCITY™ stent, both mounted on Raptor® Stent Delivery Systems. A total of 100 patients will be entered in the study and will be randomized on a 1:1 basis. Patients who meet the eligibility criteria will be either randomized to Treatment A or Treatment B. Neither the investigator nor the patient will know which stent will be implanted. Patients will be followed at 30 days, 6, 9, and 12 months, and at 2, 3, 4 and 5 years post-procedure, with all patients undergoing repeat angiography at 8 months. Additionally, medical costs associated with the index hospitalization and length of stay, and repeat hospitalizations and costs associated with other relevant medical resource use during the 5 years follow-up period will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
* Single treatment of de novo lesion in a major coronary artery in patients with single or multi-vessel disease; patients with multiple lesions can be included only if the other lesions do not require treatment;
* Target vessel diameter at the lesion site is >=2.50mm and <=3.0mm in diameter (visual estimate);
* Target lesion is >=15mm and <=32mm in length (visual estimate);
* Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

* Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
* Has unstable angina classified as Braunwald III B or C and A I-II-III, or is having a peri infarction;
* Unprotected left main coronary disease with >=50% stenosis;
* Significant (>50%) stenoses proximal or distal to the target lesion that might require revascularization or impede runoff;
* Have an ostial target lesion;
* Angiographic evidence of thrombus within target lesion;
* Heavily calcified lesion which cannot be successfully predilated;
* Documented left ventricular ejection fraction <=25%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-03; Primary Completion 2002-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
in-stent minimum lumen diameter (MLD) | 8 months

SECONDARY OUTCOMES:
composite of Major Adverse Cardiac Events defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization | 30 days and 6, 9, and 12 months, and 2, 3, 4 and 5 years
angiographic binary restenosis (³50% diameter stenosis) | 8 months
in-lesion MLD | 8 months
target lesion revascularization | 9 months
target vessel revascularization | 9 months
target vessel failure defined as cardiac death, myocardial infarction, or target vessel revascularization | 9 months
procedure success defined as achievement of a final diameter stenosis of <50% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion | up to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Erick Schampaert, MD, Principal Investigator — Hopital Sacreé-Coeur, Montréal, Canada

REFERENCES:
- [Result] Schampaert E, Cohen EA, Schluter M, Reeves F, Traboulsi M, Title LM, Kuntz RE, Popma JJ; C-SIRIUS Investigators. The Canadian study of the sirolimus-eluting stent in the treatment of patients with long de novo lesions in small native coronary arteries (C-SIRIUS). J Am Coll Cardiol. 2004 Mar 17;43(6):1110-5. doi: 10.1016/j.jacc.2004.01.024. PMID 15028375
- [Result] Rinfret S, Cohen DJ, Tahami Monfared AA, Lelorier J, Mireault J, Schampaert E. Cost effectiveness of the sirolimus-eluting stent in high-risk patients in Canada: an analysis from the C-SIRIUS trial. Am J Cardiovasc Drugs. 2006;6(3):159-68. doi: 10.2165/00129784-200606030-00003. PMID 16780389
- [Derived] Spaulding C, Daemen J, Boersma E, Cutlip DE, Serruys PW. A pooled analysis of data comparing sirolimus-eluting stents with bare-metal stents. N Engl J Med. 2007 Mar 8;356(10):989-97. doi: 10.1056/NEJMoa066633. Epub 2007 Feb 12. PMID 17296825